CLINICAL TRIAL: NCT03903419
Title: Feasibility Study for the Realization of 68Ga-PSMA PET-CT and 18F-FDOPA PET-CT for Identification of Early Recurrence in Patients Treated With Radiotherapy for Glioblastoma
Brief Title: Feasibility Study of 68Ga-PSMA PET-CT and 18F-FDOPA PET-CT in Glioblastoma's Patients
Acronym: PAraDiGM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ET18-143
Record Dates: First submitted 2019-03-28; First posted 2019-04-04 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Glioblastomas
MeSH Terms: conditions — Glioblastoma | interventions — Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA PET-CT and 18F-FDOPA PET-CT (Experimental): Functional imaging: 68Ga-PSMA and 18F-FDOPA PET-CT Immunohistochemistry of initial chirurgical sample with determination of PSMA expression
  Interventions: Diagnostic Test: Feasibility study for the realization of 68Ga-PSMA PET-CT and 18F-FDOPA PET-CT for identification of early recurrence in patients treated with radiotherapy for glioblastoma.

INTERVENTIONS:
Diagnostic Test: Feasibility study for the realization of 68Ga-PSMA PET-CT and 18F-FDOPA PET-CT for identification of early recurrence in patients treated with radiotherapy for glioblastoma. — This study is a non-randomized, prospective, feasibility study assessing 68Ga-PSMA PET-CT and 18F-FDOPA PET-CT to differentiate early recurrence from post-radiation modifications in patients treated with radiotherapy for glioblastoma.
  Patients with a MRI performed since the end of the radiotherapy until 12 months of follow up after the end of radiotherapy, will be referred for both 68Ga-PSMA and 18F-FDOPA PET-CT, whatever the conclusion of the MRI (post radiation modifications, relapse or doubtful MRI).

SUMMARY:
This study is a non-randomized, prospective, multicentric feasibility study assessing 68Ga-PSMA PET-CT and 18F-FDOPA PET-CT to differentiate early recurrence from post-radiation modifications in patients treated with radiotherapy for glioblastoma.

Patients with a MRI performed since the end of the radiotherapy until 12 months of follow up after the end of radiotherapy, will be referred for both 68Ga-PSMA and 18F-FDOPA PET-CT, whatever the conclusion of the MRI (post radiation modifications, relapse or doubtful MRI).

The rationale of doing 68Ga-PSMA and 18F-FDOPA brain PET-CT in each case will be discussed in detail with the referring physician and an informed consent will be taken from each patient for the study. The two imaging studies will be done at least with a gap of 6 hours, using the same PET-CT scanner.

DETAILED DESCRIPTION:
Gliomas are the most common primary intra-axial brain tumors arising from the glial cells. The reference treatment consists in a surgical removal followed by radiotherapy and chemotherapy (Temozolomide).

Because of frequent recurrences after first-line therapy, an accurate neuroimaging is needed. The reference anatomical modality is represented by Magnetic Resonance Imaging (MRI), especially multimodal MRI (MRI with gadolinium injection associated with spectroscopy, perfusion and diffusion). One of the particular goals of this imaging is to discriminate recurrences after therapy from radiation-related complications, which can be challenging. These last ones are side effects which turn out after radiotherapy, particularly when high doses are delivered or if chemotherapy is associated. It can occur during the first 3 months after radiotherapy as a subacute radiation related side effects and is then denominated "pseudo-progression", or after the first 3 months of completing radiotherapy as a later and chronic inflammation radiation-related complication named radiation necrosis. It can display clinical symptoms and imaging features which can mimic a relapse. Biopsy is the gold standard but may be not feasible or inconclusive due to limited and non-representative sampling.

The functional nuclear imaging usually completes the anatomical imaging in the oncological response assessment, by providing further metabolic information. Many Positron Emission Tomography (PET) tracers have been studied such as 18F-FDG exploring glucose metabolism, 18F-FLT as a nucleoside analogue, and 18F-FDOPA, 18F-FET, 11C-MET which are radiolabeled amino acids.

A new promising PET radio-tracer is currently soaring. This is the Prostate Specific Membrane Antigen (PSMA) radiolabeled with Gallium 68, a positron emitter, readily available because of a "homemade synthesis". The PSMA is a transmembrane glycoprotein over-expressed in prostate adenocarcinomas

A few studies performed glioblastomas functional imaging based on this PSMA over expression. All achieved to display glioblastomas with 68Ga-PSMA PET-scanner. A recent publication performed on five patients compared 68Ga-PSMA and 18F-FDG in the diagnostic value of glioblastomas recurrence detection. 68Ga-PSMA showed better identification of recurrent lesions owing to a higher target to background ratio. However the place of this new promising tracer in the glioblastomas monitoring remains poorly documented.

Moreover, a study reported that 18F-FDOPA was more accurate than 18F-FDG in the diagnosis of brain tumor recurrence.

To the best of our knowledge, there are no findings concerning 68GA-PSMA and 18F-FDOPA comparison in distinguishing glioblastomas recurrence from radiation-related complications.

Because of the cost and availability of 68Ga-PSMA, if its performances were better than or similar to 18F-FDOPA ones, it could tend to replace this last one in the future. Whether it could be a surrogate to the 18F-FDOPA has not been elucidated yet, representing an interesting challenge.

In this study, the investigators will evaluate the feasibility of using 68Ga-PSMA PET-CT to distinguish recurrent glioblastomas from radiation-related complications, and its comparison with 18F-FDOPA. This study will not allow a proper evaluation of the sensitivity and specificity, which will be performed in a next larger research after completion of this preliminary phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically proven glioblastoma.
* Prior treatment with radiation therapy, with or without any concomitant treatment (e.g., chemotherapy).
* MRI evaluation within the end of radiotherapy to 12 months of follow-up after the end of radiotherapy, with a diagnosis of relapse, or post radiation modifications, or doubt between tumor recurrence or radiation-related complications.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-3.
* Covered by a medical insurance.
* Signed informed consent.

Exclusion Criteria:

* Pregnancy.
* Breastfeeding.
* Adults who are subject to a protective measure or who are unable to express their consent.
* Patients treated by Avastin within 3 months.
* Patients participating in clinical trials involving isotopic ionizing imaging examinations and/or angiogenic anti-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-08-16 (Estimated); Study Completion 2021-08-16 (Estimated)

PRIMARY OUTCOMES:
Comparison of Maximum Standardized Uptake Values of 68Ga-PSMA and of 18F-FDOPA PET-CT in glioblastomas recurrences and radiation-related complications after radiotherapy. | 1 week
  Maximum Standardized Uptake Values (SUVmax) of both 68Ga-PSMA and 18F-FDOPA.
Comparison of Target to Background Ratio of 68Ga-PSMA and of 18F-FDOPA PET-CT in glioblastomas recurrences and radiation-related complications after radiotherapy. | 1 week
  Target to Background Ratio (TBR) of both 68Ga-PSMA and 18F-DOPA.
Comparison of Target to Background Ratio and Target to Striatum Ratio of 68Ga-PSMA and of 18F-FDOPA PET-CT in glioblastomas recurrences and radiation-related complications after radiotherapy. | 1 week
  Target to Background Ratio (TBR) of 68Ga-PSMA and Target to Striatum Ratio of 18F-DOPA.

SECONDARY OUTCOMES:
Description of the final diagnosis according to clinical and/or MRI follow-up. | 3 months
  Assessement of tumour recurrence or radiation-related complication.
Concordance between 68Ga-PSMA and 18F-FDOPA PET-CT from visual interpretation. | 1 week
  Measure of agreement between the two techniques using Kappa coefficient based on tracer uptake (abnormal: yes/no).
PSMA expression on initial glioblastoma sample by immunohistochemistry (IHC). | 3 months
  PSMA expression by immunohistochemistry (IHC).
Association between PSMA expression and 68Ga-PSMA PET-CT imaging data. | 3 months
  PSMA expression detectable on IHC: yes or not
Association between PSMA expression (IHC) and 68Ga- PSMA PET-CT imaging data. association between PSMA expression and 68Ga-PSMA PET-CT imaging data. | 3 months
  Measurement of PSMA uptake on PET-CT
Assessment of safety will be based mainly on the frequency of adverse events according to the common toxicity criteria (CTCAE v5.0) grade | 3 months
  The assessment of safety will be based mainly on the frequency of adverse events according to the common toxicity criteria (CTCAE v5.0) grade.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie MOREAU, M.D, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Hôpital Pierre WERTHEIMER - HCL, Bron
  - Centre Léon Berard, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McBriar JD, Shafiian N, Scharf S, Boockvar JA, Wernicke AG. Prostate-Specific Membrane Antigen Use in Glioma Management: Past, Present, and Future. Clin Nucl Med. 2024 Sep 1;49(9):806-816. doi: 10.1097/RLU.0000000000005365. Epub 2024 Jul 1. PMID 38968568